CLINICAL TRIAL: NCT06014528
Title: A Multicenter, Randomized, Double-Blind, Phase II Clinical Study of IN10018 in Combination With Pegylated Liposomal Doxorubicin (PLD) vs. Placebo in Combination With PLD for the Treatment of Platinum-resistant Recurrent Ovarian Cancer
Brief Title: IN10018 in Combination With Pegylated Liposomal Doxorubicin (PLD) vs. Placebo in Combination With PLD for the Treatment of Platinum-resistant Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN10018-011
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Intervention Model Description: Treatment allocation/randomization will be stratified according to the following factors:
  1. Prior bevacizumab use (yes or no).
  2. Platinum free interval (PFI, < 3 months or 3-6 months), 3 months is defined as 90 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind clinical study, therefore, investigator, site staff, subject, and sponsor involved in study will not know the treatment administered. In addition, the central imaging reviewer conducting the BICR evaluation will also be blinded to study treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): IN10018+PLD
  Interventions: Drug: IN10018; Drug: Pegylated Liposomal Doxorubicin
- Control Arm (Placebo Comparator): Placebo of IN10018+PLD
  Interventions: Drug: Placebo of IN10018; Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: IN10018 — 100mg QD orally (PO)
  Other Names: BI 853520
  Arms: Experimental Arm
Drug: Placebo of IN10018 — 100mg QD orally (PO)
  Arms: Control Arm
Drug: Pegylated Liposomal Doxorubicin — 40 mg/m2 once every 4 weeks (Q4W) intravenously (IV)
  Other Names: PLD

SUMMARY:
This is a multicenter, randomized, double-blind, phase II clinical study to evaluate the efficacy and safety of IN10018 in combination with PLD vs. placebo in combination with PLD in subjects with platinum-resistant recurrent ovarian cancer (including fallopian tube and primary peritoneal cancers).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, Phase II clinical study to evaluate the efficacy and safety of IN10018 in combination with PLD vs. placebo in combination with PLD in subjects with platinum-resistant recurrent ovarian cancer (including fallopian tube and primary peritoneal cancers).

Approximately 168 subjects will be enrolled into the study. Eligible subjects will be randomized in a 2: 1 ratio to receive IN10018 in combination with PLD treatment (Experimental Arm, N = approx. 112) or placebo of IN10018 in combination with PLD (Control Arm, N = approx. 56). Subjects will be stratified by prior bevacizumab use (yes or no) and platinum free interval (PFI, < 3 months or 3-6 months).

Subjects will be randomized to one of following treatment arms. The investigator should follow the clinical study protocol, the approved label of these drugs and/or institutional standard of care.

* Experimental Arm: IN10018 100 mg QD orally (PO) plus PLD 40 mg/m2 once every 4 weeks (Q4W) intravenously (IV).
* Control Arm: Placebo of IN10018 100 mg QD orally (PO) plus PLD 40 mg/m2 once every 4 weeks (Q4W) intravenously (IV).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign informed consent(s). Signed informed consent must be obtained before any study specific procedures, except those procedures used as institutional standard of care falling into the protocol specified window and fulfilling study specific requirements such as tumor imaging.
2. Female subjects ≥ 18 years at the time of signing informed consent.
3. Histologically confirmed epithelial ovarian cancer, fallopian tube cancer or primary peritoneum cancer and its subtype is high-grade serous carcinoma (HGSC).
4. Have received platinum containing therapy and have radiological relapse or progression during platinum containing treatment or < 6 months (184 calendar days) after completion of prior platinum-based therapy (at least 4 cycles).

   Note: Disease progression or recurrence requires evidence of radiographic or clinical progression (e.g., new ascites or cytological reports of pleural fluid), and elevated CA125 alone is not a criterion for progression or recurrence. Primary platinum-refractory ovarian cancers (defined as progression during or within 4 weeks after first line platinum-based therapy) is excluded, while secondary platinum-refractory disease is allowed and does not require at least 4 cycles of platinum-based therapy.
5. Maximum total of 3 prior lines of systemic therapy are allowed. Note: Hormonal therapies (e.g., tamoxifen), PARP inhibitors and bevacizumab given in the maintenance setting post response to platinum-based therapy will not count as a treatment line. Other maintenance regimens may also not count as a treatment line by discussion between the investigator and sponsor.
6. At least one measurable lesion can be accurately measured per RECIST 1.1 as assessed by investigator.

   Note: Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. ECOG performance status of 0 or 1.
8. Life expectancy of at least 3 months as assessed by investigator.
9. Availability of archival or fresh (newly obtained) tumor tissue sample during screening phase: fresh tumor tissue sample obtained after most recent relapse or progression is preferred; if no sample or not sufficient number of slides (refer to Laboratory Manual which will be provided separately) can be provided or collected, a joint decision between sponsor and investigator is needed for the enrollment of this subject.
10. Must have recovered from all AEs due to previous therapies to ≤ Grade 1 (CTCAE 5.0) or stable status as assessed by investigator.

    Note: subjects with minor toxicities with no safety concern like alopecia and Grade 2 neuropathy could be enrolled per evaluation of investigator.
11. Adequate bone marrow, liver, renal, and coagulation function within 7 days prior to randomization.

    1. Hemoglobin (Hb) ≥ 100 g/L (10 g/dL), independent of blood infusion, red blood cell transfusion and erythropoietin (EPO) use within 14 days prior to the screening period examination.
    2. Platelet count ≥ 100 × 109/L, independent of platelet infusion within 14 days prior to the screening period examination.
    3. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, independent of colony stimulating factor (CSF) use within 14 days prior to the screening period examination.
    4. Total bilirubin ≤ upper limit of normal (ULN).
    5. Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for subjects with documented liver involvement of their disease).
    6. Serum creatinine ≤ 1.5 × ULN, Estimated Creatinine clearance rate (Clcr) by the Cockcroft-Gault (C-G) equation ≥ 60 mL/min or estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) equation ≥ 60 mL/min.
    7. Urinary protein negative or trace (±); or urinary protein ≥ 1+ but with a urine protein to creatinine ratio (UPCR) in a morning spot urine sample < 0.5 or a 24-hour urine protein < 0.5 g/24 h.
    8. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Subjects with stable anticoagulation treatment is allowed.
12. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in section 10.4 Appendix 4 of the full protocol.

       OR
    2. A WOCBP who agrees to follow the contraceptive guidance in section 10.4 Appendix 4 of the full protocol during the treatment period and through 3 months after the last dose of study treatment.

Exclusion Criteria:

1. Has had major surgery or significant traumatic injury within 28 days prior to randomization, or diagnostic biopsies within 14 days prior to randomization.

   Note: Subjects with anticipation of the need for major surgery during study treatment should be excluded. Subjects who underwent diagnostic biopsy within 14 days prior to randomization may also be enrolled if the investigator and sponsor determine that the diagnostic biopsy will not affect the efficacy evaluation.
2. Has received prior systemic anticancer therapy including investigational agents, such as within 14 days or less than 5 half-lives (whichever is shorter) of chemotherapy or targeted therapy, or within 28 days of immunotherapy, macromolecular drugs (eg., bevacizumab) or investigational drugs prior to randomization.
3. Has received prior radiotherapy within 14 days prior to randomization. Note: A 7-day washout is permitted for palliative radiation (≤ 14 days of radiotherapy) to non-central nervous system (CNS) disease.
4. Has received prior treatment of any FAK inhibitor or prior treatment of PLD.
5. Has a known previous or concurrent cancer that is distinct in primary site or histology from current ovarian cancer within 3 years prior to randomization, except for curatively treated cancers such as cervical/breast/prostate carcinoma in situ and basal cell carcinoma.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Subjects with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression) for at least 4 weeks apart by repeat imaging (note that the repeat imaging should be performed during screening phase) for at least 28 days prior to randomization.
7. Has a history of major cardiovascular, cerebrovascular or thromboembolic diseases (e.g., congestive heart failure, acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism) within 6 months before randomization, or has any of the following abnormality:

   1. QTc interval corrected using Fridericia's formula > 470 ms (based on QTcF).
   2. Left ventricular ejection fraction (LVEF) < 50%.
   3. New York Heart Association (NYHA) functional classification ≥ Grade 2.
   4. Clinically significant arrhythmia.
   5. Uncontrolled hypertension or diabetes.
   6. Other clinically significant heart diseases.
8. Has known pleural effusion, pericardial effusion or ascites accompanied by clinical symptoms or requiring puncture or drainage. Subjects who received drainage within the first 3 months of randomization should be excluded. A small amount of ascites that can only be detected by imaging examination and without clinical symptom is allowed.
9. Has malabsorption syndrome or inability to take oral drugs.
10. Has clinically significant gastrointestinal abnormalities including uncontrolled gastrointestinal inflammatory lesions (Crohn's disease, or ulcerative colitis in active) or uncontrolled gastrointestinal bleeding.
11. Clinical or radiographic evidence of intestinal obstruction, or aetiology of previous recurrent ileus not excluded.
12. Currently have interstitial pneumonia (except for radiation pulmonary fibrosis that does not require hormonal therapy).
13. Has not well controlled active infection after systemic therapy.
14. Has known human immunodeficiency virus (HIV) infection or known active Hepatitis B or Hepatitis C virus infection.

    Note: No HIV, Hepatitis B and Hepatitis C testing is required unless mandated by local health authority and/or site.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
17. Known allergy or hypersensitivity to IN10018 or PLD, or their ingredients.
18. Has received prior cumulative anthracycline dose of 550 mg/m2 or more.
19. Has received systemic treatment of CYP3A4, CYP2D6 or P-gp strong inhibitors/inducers within 14 days prior to randomization, or anticipation of the systemic treatment of these drugs during Treatment Phase.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per RECIST 1.1, as assessed by blinded independent central review (BICR), following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  PFS per RECIST 1.1, as assessed by BICR.

SECONDARY OUTCOMES:
Overall survival (OS), following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 3 years.
  OS
Progression-free survival (PFS) per RECIST 1.1, as assessed by investigator , following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  Defined as the proportion of subjects with complete response (CR) or partial response (PR)
Objective response rate (ORR) per RECIST 1.1, as assessed by BICR and Investigator, following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  Defined as the proportion of subjects with complete response (CR) or partial response (PR)
Disease control rate (DCR) per RECIST 1.1, as assessed by BICR and Investigator, following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
Duration of response (DoR) per RECIST 1.1, as assessed by BICR and Investigator, following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
Safety and tolerability of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  The number of participants who experienced AEs is presented.

OTHER OUTCOMES:
CA 125 response rate per Gynecological Cancer Intergroup (GCIG) criteria, following treatment of IN10018 in combination with PLD vs. placebo in combination with PLD. | 2 years.
  CA 125 response rate per GCIG criteria.
PK: AUC0-τ of subjects receiving IN10018 and/or PLD treatment by serial and sparse PK samplings. | 2 years.
  Area under the concentration-time curve (AUC)
PK: Ctrough of subjects receiving IN10018 and/or PLD treatment by serial and sparse PK samplings. | 2 years.
  Trough concentration (Ctrough)
PK: Cmax of subjects receiving IN10018 and/or PLD treatment by serial and sparse PK samplings. | 2 years.
  PK parameters (i.e., AUC0-τ, Cmax and Ctrough) of IN10018 and PLD, and expose-response relationship of IN10018 by population PK models.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying WU, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China